CLINICAL TRIAL: NCT02555709
Title: A Randomized, Double-Blind, Placebo-Controlled Ascending Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VTP-43742 in Healthy Volunteers and Psoriatic Patients and Clinical Proof-of-Concept in Psoriatic Patients
Brief Title: An Ascending Multiple Dose Study With VTP-43742 in Healthy Volunteers and Psoriatic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vitae Pharmaceuticals Inc., an Allergan affiliate (Industry)
Responsible Party: Sponsor
Organization: Vitae Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: VTP-43742-002
Record Dates: First submitted 2015-09-15; First posted 2015-09-21 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — VTP-43742

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (13):
- Placebo 1 (Placebo Comparator): healthy volunteers
  Interventions: Drug: Placebo 1
- VTP-43742 Dose 1 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 2 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 3 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 4 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 5 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 6 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 7 (Experimental): healthy volunteers
  Interventions: Drug: VTP-43742
- Placebo 2 (Placebo Comparator): psoriatic patients
  Interventions: Drug: Placebo 2
- VTP-43742 Dose 8 (Experimental): psoriatic patients
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 9 (Experimental): psoriatic patients
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 10 (Experimental): psoriatic patients
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 11 (Experimental): psoriatic patients
  Interventions: Drug: VTP-43742

INTERVENTIONS:
Drug: VTP-43742 — VTP-43742 administered as an oral capsule once daily
  Arms: VTP-43742 Dose 1; VTP-43742 Dose 10; VTP-43742 Dose 11; VTP-43742 Dose 2; VTP-43742 Dose 3; VTP-43742 Dose 4; VTP-43742 Dose 5; VTP-43742 Dose 6; VTP-43742 Dose 7; VTP-43742 Dose 8; VTP-43742 Dose 9
Drug: Placebo 1 — Placebo 1 matching VTP-43742 administered as an oral capsule once daily
  Arms: Placebo 1
Drug: Placebo 2 — Placebo 2 matching VTP-43742 administered as an oral capsule once daily
  Arms: Placebo 2

SUMMARY:
This is a two-part, randomized, double-blind, placebo-controlled study in which VTP-43742 will be administered to normal healthy volunteers (NHV) and to moderate to severe psoriatic patients, both in sequential ascending dose panels.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled, ascending multiple dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics effects of VTP-43742 in healthy volunteers conducted at a single, study center and in patients with moderate to severe chronic plaque-type psoriasis at approximately 8 study centers in the United States. A total of 108 participants will be enrolled in the study (48 healthy subjects and 60 psoriatic patients).

ELIGIBILITY:
Healthy Volunteer Inclusion Criteria:

* Healthy males or females, 18 to 45 years of age, inclusive.
* Body weight of at least 55 kg and body mass index of 18-32 kg/m2, inclusive.
* Medically healthy with clinically insignificant screening results.
* Women of child-bearing potential (WOCBP) may be enrolled if they agree to use two of the reliable forms of contraception
* Men with partners who are WOCBP must agree that they and/or their partner will use two of the reliable forms of contraception
* WOCBP must have a negative serum βhCG pregnancy test at the Check-in visit.
* Voluntarily consent to participate in the trial

Psoriasis Patient Inclusion Criteria:

* Confirmed diagnosis of chronic plaque-type psoriasis, diagnosed at least 6 months before study with at least moderate severity, which is defined as PASI≥10, PGA≥3, and % BSA≥8
* Otherwise medically healthy and with otherwise clinically insignificant screening laboratory test results
* Males or females, 18 to 75 years of age, inclusive
* Body weight of at least 55 kg and body mass index of 18-35 kg/m2, inclusive.
* WOCBP may be enrolled if they agree to use two of the reliable forms of contraception
* Men with partners who are WOCBP must agree that they and/or their partner will use two of the reliable forms of contraception
* WOCBP must have a negative serum β hCG pregnancy test at the Screening and Baseline visit
* Voluntarily consent to participate in the trial

Healthy Volunteer Exclusion Criteria:

* Unwilling or unable to provide written informed consent
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, coagulation, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Evidence of organ dysfunction or any clinically significant deviation from normal in vital signs, physical examination, clinical laboratory determinations or ECG
* Any major surgery within 3 months of Screening
* Positive urine drug/alcohol testing at Screening or Baseline visit
* Use of tobacco and/or nicotine-containing products within 3 months prior to the start of dosing of the trial
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV Ab) at Screening
* History or presence of alcoholism or drug abuse as defined in DSM V, Diagnostic Criteria for Drug and Alcohol Abuse
* History of hypersensitivity or idiosyncratic reaction to drugs from multiple drug classes
* Any previous gastrointestinal surgery or recent (within 3 months) history of gastrointestinal disease that could impact the absorption of the study drug
* Blood donation or significant blood loss within 8 weeks prior to Day 1of the trial
* Plasma donation within 7 days prior to Day 1 of the trial
* Blood transfusion within 4 weeks of Screening
* Positive serum pregnancy test (WOCBP) at the Screening or Baseline visit
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical disease (e.g., infectious disease) must not be enrolled into this study
* Any other medical, psychiatric, and /or social reason as determined by the Investigator

Psoriatic Patient Exclusion Criteria:

* Unwilling or unable to provide written informed consent
* Efficacy failure on two or more biological agents for the treatment of psoriasis when the failures occurred within one year of the initiation of the therapy of the first biological agent
* Current treatment or history of treatment for psoriasis with biologicals within 6 months of study Day 1
* Current treatment or history of treatment for psoriasis with non-biological systemic medications within 4 weeks of Day 1 and treatment with topical agents within 2 weeks of Day 1
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, coagulation, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Evidence of organ dysfunction or any clinically significant deviation from normal in vital signs, physical examination, clinical laboratory determinations or ECG
* Any major surgery within 3 months of Screening
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV Ab) at Screening
* History or presence of alcoholism or drug abuse as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse
* History of hypersensitivity or idiosyncratic reaction to drugs from multiple drug classes
* Any previous gastrointestinal surgery or recent (within 3 months) history of gastrointestinal disease that could impact the absorption of the study drug
* Blood donation or significant blood loss within 8 weeks prior to Day 1 of the trial
* Plasma donation within 7 days prior to Day 1 of the trial
* Blood transfusion within 4 weeks of Screening
* Positive serum pregnancy test (WOCBP) at the Screening or positive urine pregnancy test with confirmatory serum pregnancy test on Day 1
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical disease (e.g., infectious disease) must not be enrolled into this study.
* Any other medical, psychiatric, and /or social reason as determined by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
safety data, including AEs, laboratory evaluations, ECG results, and vital signs assessments, will be listed by subject and summarized by dose and time point | 10 days
safety data, including AEs, laboratory evaluations, ECG results, and vital signs assessments, will be listed by subject and summarized by dose and time point | 28 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) will be summarized using descriptive statistics by visit and dose level | Day 1, 10 and 28
Time to maximum plasma concentrations (tmax) will be summarized using descriptive statistics by visit and dose level | Day 1, 10 and 28
The area under the plasma concentration versus time curve, from time 0 to the last measurable concentration (AUCt) will be summarized using descriptive statistics by visit and dose level | Day 1, 10 and 28
The area under the plasma concentration versus time curve, from time 0 to infinity (by extrapolation) (AUC∞) will be summarized using descriptive statistics by visit and dose level | Day 1, 10 and 28
Half life (t½) will be summarized using descriptive statistics by visit and dose level | Day 1, 10 and 28
Percent change from baseline in total PASI will be summarized using descriptive statistics by visit and dose level | 28 days

OTHER OUTCOMES:
changes from baseline and/or placebo for IL-17 plasma levels | Day 1, 10 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gregg, MD, Study Director — Vitae Pharmaceuticals
Locations (14):
- United States (14):
  - Patient Site 5, Rogers, Arkansas
  - Patient Site 1, Miami, Florida
  - Patient Site 8, Tampa, Florida
  - Patient 12, Tampa, Florida
  - Patient Site 13, Carmel, Indiana
  - Patient Site 4, Plainfield, Indiana
  - Healthy Volunteer Site 1, Fair Lawn, New Jersey
  - Patient Site 2, New York, New York
  - Patient Site 9, High Point, North Carolina
  - Patient Site 6, College Station, Texas
  - Patient Site 3, Dallas, Texas
  - Patient Site 10, Houston, Texas
  - Patient Site 11, Houston, Texas
  - Patient Site 7, Webster, Texas